CLINICAL TRIAL: NCT03205943
Title: Use of a Non-invasive Bio-impedance Cardiac Monitor, ICON™, to Detect and Trend Hemodynamic Variables During Dexmedetomidine Sedation in Children Undergoing Pulmonary Function Testing
Brief Title: Use of ICON™ to Detect Hemodynamic Variables During Dexmedetomidine Sedation in Children Undergoing Pulmonary Function Test
Status: Withdrawn | Type: Observational
Why Stopped: logistical challenges
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Keira Mason, Director, Radiology Anesthesia; Senior Associate in Perioperative Anesthesia, Associate Professor of Anaesthesia, Boston Children's Hospital
Other Study IDs: P00008608
Record Dates: First submitted 2015-07-28; First posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Inadequate; Pulmonary Function, Newborn
Keywords: ICON

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To collect and analyze the physiologic data of the ICON™ during dexmedetomidine (DEX) sedation for neonatal pulmonary function testing. The ICON™ is a noninvasive physiological monitor which uses respiratory impedance to follow systemic vascular resistance (SVR), heart rate, cardiac index and stroke index.

DETAILED DESCRIPTION:
Traditionally the measurements of cardiac indices and hemodynamic variables require invasive monitors such as pulmonary thermodilution catheters and transesophageal Doppler echocardiography. In recent years, electrical cardiometry has been used for the non-invasive determination of stroke volume, cardiac output, and other hemodynamic parameters in adults, children, and neonates. Electrical cardiometry has been validated against "gold standard" methods such as thermodilution and is a proprietary method trademarked by Cardiotronic, Inc. (La Jolla, CA). Cardiotronic markets the ICON™. It is FDA-approved for use in pediatric and adult patients, is currently used for clinical purposes in the BCH MSICU at 11 South.

The ICON™ is a comprehensive, standalone hemodynamic monitor, which provides a complete hemodynamic monitoring system that provides user-defined hemodynamic parameters. It provides a continuous trend of cardiac output and stroke volume associated with rapid changes in vital signs with minimal risk to the patient.

The ICON™ monitor has been used in Boston Children's Hospital to determine the hemodynamic changes in children aged 1 month to 18 years of age who received dexmedetomidine sedation for CT and Nuclear Medicine.

Dexmedetomidine (DEX) has been found to be an effective drug in the pediatric population in both the intensive care unit and for procedures in Radiology. In a recent study, DEX caused bradycardia (3%), hypotension (9%) and hypertension (8%) in pediatric critical care patients. Intravenously administrated sedation. DEX will be delivered as per the DEX order set used for non-painful procedures in the radiology department. As an alpha 2 adrenergic agonist, DEX produces hemodynamic changes to blood pressure and heart rate. To precisely follow the trend of complex changes in systemic vascular resistance, cardiac output and stroke volume during DEX administration, would ideally be with invasive intravascular monitors which would not be warranted in pediatric sedation procedures. However, a minimal risk non-invasive cardiac output monitor such as the ICON can measure, detect, and trend these physiological changes in the neonates and infants who are receiving DEX for pulmonary function tests.

Children with certain lung conditions undergo pulmonary function tests (PFT) which are currently being performed using chloral hydrate administered by the responsible and sedation credentialed pulmonologist (Dr. Lawrence Rhein). Chloral hydrate is inconsistent and unreliable in producing adequate sedation for a successful PFT study. Sedation physicians from the BCH Department of Anesthesia have agreed to provide sedation for these patients with dexmedetomidine (DEX), using the same approved protocols that are being used in the BCH Department of Radiology for non-painful imaging studies.

Investigators will use the ICON™ to follow the physiological cardiac parameters (non-invasive blood pressure, pulse oximeter, capnography, heart rate, and electrocardiogram) throughout the pre-sedation, sedation and recovery period. Investigators propose collecting this data in a prospective manner with parental informed consent for the data collection.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 1-18 months of age, scheduled for pulmonary function testing and eligible for sedation with dexmedetomidine and whose family agree to participate in the study

Exclusion Criteria:

* Patients with the following diagnoses are not medically appropriate to receive nursing administered sedation with dexmedetomidine:
* Active, uncontrolled gastroesophageal reflux - an aspiration risk
* Active, uncontrolled vomiting - an aspiration risk
* Current (or within past 3 months) history of apnea requiring an apnea monitor
* Active, current respiratory issues that are different from the baseline status (pneumonia, exacerbation of asthma, bronchiolitis, respiratory syncytial virus)
* Unstable cardiac status (life threatening arrhythmias, abnormal cardiac anatomy, significant cardiac dysfunction)
* Craniofacial anomaly, which could make it difficult to effectively establish a mask airway for positive pressure ventilation if needed
* History of digoxin use
* Moya-Moya disease
* New-onset stroke

In addition, the following are contraindications to the use of the ICON™:

* Pacemakers
* Mitral or aorta valve dysfunction
* Dextrocardia
* Second or third degree heart block
* Current diagnosis of cardiac, pulmonary, hepatic or renal failure
* Current diagnosis of pulmonary masses/tumor/pleural effusions/pneumonia/edema
* Pericardial effusion
* Large implanted thoracic metallic devices (including orthodontic braces, spine rods, plates and screws)
* Allergy to device standard BCH ECG electrodes (Vermed A 10061-SRT disposable prewired medical electrodes)

Ages: 1 Month to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients 1-18 months, undergoing pulmonary function testing
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-12 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Changes in heart rate | Up to 12 hours
  The changes in heart rate from baseline, during the DEX administration and sedation and during recovery period (following discontinuation of the DEX) through time of discharge.
Changes in blood pressure | Up to 12 hours
  The changes in blood pressure from baseline, during the DEX administration and sedation and during recovery period (following discontinuation of the DEX) through time of discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Keira Mason, MD, Principal Investigator — Boston Children's Hospital

REFERENCES:
- [Background] Snapir A, Posti J, Kentala E, Koskenvuo J, Sundell J, Tuunanen H, Hakala K, Scheinin H, Knuuti J, Scheinin M. Effects of low and high plasma concentrations of dexmedetomidine on myocardial perfusion and cardiac function in healthy male subjects. Anesthesiology. 2006 Nov;105(5):902-10; quiz 1069-70. doi: 10.1097/00000542-200611000-00010. PMID 17065883
- [Background] Wong J, Steil GM, Curtis M, Papas A, Zurakowski D, Mason KP. Cardiovascular effects of dexmedetomidine sedation in children. Anesth Analg. 2012 Jan;114(1):193-9. doi: 10.1213/ANE.0b013e3182326d5a. Epub 2011 Sep 29. PMID 21965374